CLINICAL TRIAL: NCT03471624
Title: Treatment Outcomes in Chronic Hepatitis B Patients on Sequential Therapy With Tenofovir Alafenamide (TAF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Mindie H. Nguyen, Profesor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 45054
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hepatitis B, Chronic
Keywords: Tenofovir alafenamide (TAF)
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tenofovir Alafenamide for 24 months (Experimental): Participants on any antiviral treatment for chronic HBV who plan to be switched by their physician to be treated with TAF 25 mg for 24 months.
  Interventions: Drug: Tenofovir Alafenamide

INTERVENTIONS:
Drug: Tenofovir Alafenamide — Tenofovir alafenamide (TAF) is a new formulation of tenofovir with higher intracellular active drug concentration allowing for dosing of only 25 mg once daily and thus can potentially lower the already low risk of renal toxicity and bone loss with tenofovir disoproxil fumarate (TDF).
  Other Names: Vemlidy

SUMMARY:
Primary Objective:

To describe rate of persistence and/or improvement of viral suppression with TAF as with previous anti-HBV (hepatitis B virus) treatment

DETAILED DESCRIPTION:
Secondary Objective(s):

1. Describe persistence of ALT (alanine aminotransferase) normalization and/or improvement of ALT levels with TAF as with previous anti-HBV treatment
2. To describe trends in serum creatinine and calculated creatinine clearance as available by local labs.
3. To describe trends in bone mass from baseline to 24 months after switch.

https://med.stanford.edu/nguyenlab/clinical-trials.html

ELIGIBILITY:
Inclusion criteria:

1. Male or female, age ≥18 years
2. Chronic hepatitis B diagnosis confirmed by positive HBsAg or HBV DNA or HBeAg or documented history of chronic hepatitis B in physician note
3. Currently maintained on antiviral therapy for at least 48 weeks with any Hepatitis B virus(HBV) DNA value at Screening/Baseline and planned to be switched to TAF by their physician
4. Routinely monitored for serum HBV DNA Polymerase chain reaction(PCR), liver chemistry including Aspartate aminotransferase (AST )/alanine transaminase(ALT)/total bilirubin, renal chemistry including Blood urea nitrogen(BUN)/Creatinine/Carbon dioxide (CO2) by their physicians every 3-6 months and a bone density scan at least every 2 years as per routine clinical care (one at baseline and one 2 years after switch).
5. Estimated creatinine clearance > 15 ml/min (using the Cockcroft-Gault method) at Screening/Baseline Visit. (Note: multiply estimated rate by 0.85 for women).
6. Willing and able to provide informed consent
7. Able to comply with dosing instructions for study drug administration and able to complete the study schedule of assessments

Exclusion criteria:

1. Pregnant women, women who are breastfeeding or who believe they may wish to become pregnant during the course of the study
2. Previous recipient of a liver transplant
3. Co-infection with human immunodeficiency virus (HIV) or hepatitis C (HCV) or hepatitis D (HDV)
4. Severe or uncontrolled comorbidities
5. Current or known hepatic decompensation (≤2 years) (e.g ascites, encephalopathy, or variceal hemorrhage) with a Child-Pugh score of B or C
6. Malignancy including liver cancer within 5 years except cancers curable by surgical resection (e.g. basal cell skin cancer and squamous cell cancer)
7. On any of the disallowed concomitant medications listed in the prior and concomitant medications list (pg. 11). Subjects on prohibited medications who are otherwise eligible will need a wash out period of at least 30 days prior to the Screening/Baseline visit.
8. Males and females of reproductive potential who are unwilling to use "effective" protocol-specified method(s) of contraception during the study.
9. Current substance or alcohol abuse judged by the investigator to potentially interfere with subject compliance.
10. Any other clinical conditions that, in the opinion of the Investigator, would make the subject unsuitable or unable to comply with any of the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mindie H Nguyen, MD,MAS, Principal Investigator — Stanford University
Locations (12):
- United States (2):
  - Stanford University Medical Center, Palo Alto, California
  - San Jose Gastroenterology, San Jose, California
- Japan (4):
  - Kyushu University Hospital, Fukuoka
  - Nagoya City University, Nagoya
  - Osaka City University, Osaka
  - Saga University Hospital, Saga
- South Korea (3):
  - Hanyang University Seoul Hospital, Seoul
  - Nowon Eulji Medical Center, Eulji University College of Medicine,, Seoul
  - Sanggye Paik Hospital, Inje University College of Medicine, Seoul
- Taiwan (3):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung

REFERENCES:
- [Background] Martin P, Lau DT, Nguyen MH, Janssen HL, Dieterich DT, Peters MG, Jacobson IM. A Treatment Algorithm for the Management of Chronic Hepatitis B Virus Infection in the United States: 2015 Update. Clin Gastroenterol Hepatol. 2015 Nov;13(12):2071-87.e16. doi: 10.1016/j.cgh.2015.07.007. Epub 2015 Jul 15. PMID 26188135
- [Background] Lok AS, McMahon BJ, Brown RS Jr, Wong JB, Ahmed AT, Farah W, Almasri J, Alahdab F, Benkhadra K, Mouchli MA, Singh S, Mohamed EA, Abu Dabrh AM, Prokop LJ, Wang Z, Murad MH, Mohammed K. Antiviral therapy for chronic hepatitis B viral infection in adults: A systematic review and meta-analysis. Hepatology. 2016 Jan;63(1):284-306. doi: 10.1002/hep.28280. Epub 2015 Nov 13. PMID 26566246
- [Background] Schweitzer A, Horn J, Mikolajczyk RT, Krause G, Ott JJ. Estimations of worldwide prevalence of chronic hepatitis B virus infection: a systematic review of data published between 1965 and 2013. Lancet. 2015 Oct 17;386(10003):1546-55. doi: 10.1016/S0140-6736(15)61412-X. Epub 2015 Jul 28. PMID 26231459
- [Background] Weinbaum CM, Williams I, Mast EE, Wang SA, Finelli L, Wasley A, Neitzel SM, Ward JW; Centers for Disease Control and Prevention (CDC). Recommendations for identification and public health management of persons with chronic hepatitis B virus infection. MMWR Recomm Rep. 2008 Sep 19;57(RR-8):1-20. PMID 18802412
- [Background] Ward JW, Byrd KK. Hepatitis B in the United States: a major health disparity affecting many foreign-born populations. Hepatology. 2012 Aug;56(2):419-21. doi: 10.1002/hep.25799. No abstract available. PMID 22532028
- [Background] Sarin SK, Kumar M, Lau GK, Abbas Z, Chan HL, Chen CJ, Chen DS, Chen HL, Chen PJ, Chien RN, Dokmeci AK, Gane E, Hou JL, Jafri W, Jia J, Kim JH, Lai CL, Lee HC, Lim SG, Liu CJ, Locarnini S, Al Mahtab M, Mohamed R, Omata M, Park J, Piratvisuth T, Sharma BC, Sollano J, Wang FS, Wei L, Yuen MF, Zheng SS, Kao JH. Asian-Pacific clinical practice guidelines on the management of hepatitis B: a 2015 update. Hepatol Int. 2016 Jan;10(1):1-98. doi: 10.1007/s12072-015-9675-4. Epub 2015 Nov 13. PMID 26563120
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Result] Ogawa E, Jun DW, Toyoda H, Hsu YC, Yoon EL, Ahn SB, Yeh ML, Do S, Trinh HN, Takahashi H, Enomoto M, Kawada N, Yasuda S, Tseng CH, Kawashima K, Lee HA, Inoue K, Haga H, Do AT, Maeda M, Hoang JH, Cheung R, Ueno Y, Eguchi Y, Furusyo N, Yu ML, Tanaka Y, Nguyen MH. Increased spine bone density in patients with chronic hepatitis B switched to tenofovir alafenamide: A prospective, multinational study. Aliment Pharmacol Ther. 2024 Jan;59(2):239-248. doi: 10.1111/apt.17785. Epub 2023 Oct 26. PMID 37882252
- See also: Vemlidy package insert — https://www.gilead.com/~/media/files/pdfs/medicines/liver-disease/vemlidy/vemlidy_pi.pdf?la=en

RESULTS

PARTICIPANT FLOW:
Groups:
- Tenofovir Alafenamide for 24 Months: Participants with chronic hepatitis B virus (HBV) infection receive tenofovir alafenamide (TAF) 25 mg for 24 months.
Period: Overall Study
Arm/Group | Tenofovir Alafenamide for 24 Months
Started | 270
Completed | 258
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: 270 completed study enrollment procedures and were included in study analysis
Groups:
- Tenofovir Alafenamide for 24 Months: Participants with chronic HBV infection receive TAF 25 mg for 24 months.
Arm/Group | Tenofovir Alafenamide for 24 Months
Number analyzed (Participants) | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 187
  >=65 years | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 269
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 269
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 63
  United States | 31
  Japan | 123
  Taiwan | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HBV DNA <20 IU Per mL
Description: To describe rate of persistence and/or improvement of viral suppression with TAF as with previous anti-HBV treatment.
Time Frame: Baseline, 6, 12, 18, 24 months
Population: Participants with data at each respective time point are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Alafenamide for 24 Months
Number analyzed (Participants) | 270
Participants
  Baseline | 257
  month 6: number analyzed (Participants) | 265
  month 6 | 261
  month 12: number analyzed (Participants) | 262
  month 12 | 257
  month 18: number analyzed (Participants) | 259
  month 18 | 256
  month 24: number analyzed (Participants) | 258
  month 24 | 255

2. Secondary Outcome: Number of Participants With Normal Alanine Aminotransferase (ALT).
Description: Alanine aminotransferase (ALT) normalization is defined if ALT was less than 35 U/L for men or 25 U/L for women
Time Frame: Baseline, 6, 12, 18, 24 months
Population: Participants with data at each respective time point are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Alafenamide for 24 Months
Number analyzed (Participants) | 270
Participants
  Baseline | 203
  month 6: number analyzed (Participants) | 265
  month 6 | 212
  month 12: number analyzed (Participants) | 262
  month 12 | 197
  month 18: number analyzed (Participants) | 259
  month 18 | 203
  month 24: number analyzed (Participants) | 258
  month 24 | 203

3. Secondary Outcome: Calculated eGFR
Description: To describe trends in calculated eGFR as available by local labs. Estimated glomerular filtration rates (eGFR) were calculated using the Chronic Kidney Disease Epidemiology Collaboration(CKD-EPI) equation (eGFR [mL∕min∕1.73m2] =141 × [minimum Scr∕K, 1]α × [maximum Scr/K, 1]1.209 × 0.993age × 1.018 [if female] × 1.159 [if black]) where Scr is serum creatinine in µmol/L, K is 61.9 for females and 79.6 for males, α is -0.329 for females and -0.411 for males
Time Frame: Baseline, 6, 12, 18, 24 months
Population: Participants with data at each respective time point are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73m^2
Arm/Group | Tenofovir Alafenamide for 24 Months
Number analyzed (Participants) | 270
mL/min/1.73m^2
  Baseline | 90.2 [79.0 to 99.8]
  month 6: number analyzed (Participants) | 265
  month 6 | 90.8 [76.9 to 100]
  month 12: number analyzed (Participants) | 262
  month 12 | 91.2 [78 to 101.1]
  month 18: number analyzed (Participants) | 259
  month 18 | 91.8 [79.9 to 101.7]
  month 24: number analyzed (Participants) | 258
  month 24 | 92.1 [78.8 to 101.0]

4. Secondary Outcome: The Mean Bone Mass Density (T-score) Change
Description: To describe trends in bone mass density from baseline to end of study. Bone Mass Density(BMD) was evaluated using T-score of Lumber-spine. The T-score is a comparison of the results to a average peak bone mass of healthy young adult. 0 indicates healthy young adult's mean with a SD of 1. Normal BMD was defined with T-score of -1.0 or above; osteopenia with T-score between -1.1 and -2.4, and osteoporosis with T-score of -2.5 or below (ref). Worsened BMD was defined by upstaging of BMD class from normal to osteopenia or worse or from osteopenia to osteoporosis. Improved BMD was defined by downstaging of BMD class from osteopenia to normal or osteoporosis to osteopenia or normal.
Time Frame: Baseline, month 24
Population: Participants with data at each respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Tenofovir Alafenamide for 24 Months
Number analyzed (Participants) | 270
T-score
  Baseline | -1.43 (1.36)
  24 month: number analyzed (Participants) | 258
  24 month | -1.17 (1.38)

ADVERSE EVENTS:
Time Frame: Up to 24 months
Arm/Group | Tenofovir Alafenamide for 24 Months
All-Cause Mortality (participants affected / at risk) | 1/270
Serious Adverse Events (participants affected / at risk) | 15/270
Other Adverse Events (participants affected / at risk) | 4/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir Alafenamide for 24 Months (N=270)
Gallbladder carcinoma (Hepatobiliary disorders) | 1 (1)
Hepatocellular carcinoma (Hepatobiliary disorders) | 4 (4)
Non-Hodgkin's Lymphoma (Blood and lymphatic system disorders) | 1 (1)
Skin T cell Lymphoma (Skin and subcutaneous tissue disorders) | 1 (1)
Prostate cancer (Reproductive system and breast disorders) | 1 (1)
Breast cancer (Reproductive system and breast disorders) | 1 (1)
Rectal adenocarcinoma (Gastrointestinal disorders) | 1 (1)
Myelodysplastic syndrome (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Brain hemorrhage (Nervous system disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Left Knee osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir Alafenamide for 24 Months (N=270)
Nausea (Gastrointestinal disorders) | 3 (3)
Body pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT03471624/Prot_SAP_000.pdf